CLINICAL TRIAL: NCT04532801
Title: Evaluation of Kisspeptin Glucose-Stimulated Insulin Secretion With Physiologic Mixed Meal Tolerance
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Interim analysis of data collected under other clinical trials demonstrated planned enrollment was insufficiently powered.
Sponsor: Stephanie B. Seminara, MD (Other)
Responsible Party: Sponsor-Investigator, Stephanie B. Seminara, MD, Chief, Reproductive Endocrine Unit; Professor of Medicine, Harvard Medical School; Director, Harvard Reproductive Endocrine Sciences Center, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 267337
Record Dates: First submitted 2020-08-23; First posted 2020-08-31 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Insulin; Glucose; Healthy Volunteers; Women; Pregnancy
Keywords: kisspeptin; follicular phase
MeSH Terms: conditions — Insulin Resistance | interventions — KISS1 protein, human; Kisspeptins

STUDY DESIGN:
Intervention Model Description: physiologic studies
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- kisspeptin-10 (Experimental): kisspeptin infusion
  Interventions: Drug: Kisspeptin-10; Other: mixed meal tolerance test
- placebo (Placebo Comparator): placebo
  Interventions: Other: mixed meal tolerance test

INTERVENTIONS:
Drug: Kisspeptin-10 — kisspeptin-10 IV infusion
  Other Names: kisspeptin
  Arms: kisspeptin-10
Other: mixed meal tolerance test — mixed meal tolerance test

SUMMARY:
This study utilizes infusions of kisspeptin in healthy women to isolate the impact of kisspeptin on beta-cell responsivity assessed by the mixed meal tolerance test.

DETAILED DESCRIPTION:
Assignment: each study subject serves as their own control, and will come in timed to their cycle. The order in which they undergo the kisspeptin or placebo arms is randomized and separated by greater than two weeks to minimize variability and study-specific effects.

Delivery of Interventions:

Prior to each visit, study subjects will be asked to:

* eat at least 150 gm carbohydrates per day
* refrain from strenuous exercise

On the day of the visit, study subjects will:

* eat a standardized meal prepared by the metabolic kitchen in the clinical research center
* be observed overnight to ensure a 12-hour fast
* have an IV placed, for a 16 hour kisspeptin or placebo infusion
* after the 12 hour fast, starting at 8 am in the morning will undergo a mixed meal tolerance test

ELIGIBILITY:
HISTORY

* no personal history of chronic disease, except well controlled thyroid disease
* no history of diabetes in a first degree relative, including gestational diabetes
* no family or personal history of hyperlipidemia
* normal timing of menarche (age 10-14)
* normal menstrual cycles (q25-35 days)
* no use of contraceptive pills, patches or vaginal rings within last 4 weeks
* nulliparous (no history of a pregnancy)
* no active illicit drug use
* no history of a medication reaction requiring emergency medical care
* no difficulty with blood draws
* stable weight for previous three months
* available for all parts of the study

PHYSICAL

* body mass index (18.5-25)
* systolic BP < 120mm Hg, diastolic < 80 mm Hg
* normal waist circumference (less than 32 inches)

LABORATORY STUDIES: (per Massachusetts General Hospital reference ranges)

* fasting LDL cholesterol less than 130 mg/dL
* fasting triglycerides less than 150 mg/dL
* normal hemoglobin
* hemoglobin A1C < 5.7%
* blood urea nitrogen, creatinine not elevated
* AST, ALT not elevated
* negative serum pregnancy test

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-21 (Estimated)

PRIMARY OUTCOMES:
Beta-cell responsivity index | up to 6 months
  Average beta-cell responsivity index derived from mixed meal tolerance data comparing placebo and kisspeptin arms

OTHER OUTCOMES:
Fasting insulin level | up to 6 months
  Average fasting insulin level comparing placebo and kisspeptin arms

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Lippincott, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No